CLINICAL TRIAL: NCT06819176
Title: Lenacapavir Intensification to Disrupt HIV Reservoirs in Virologically Suppressed People With HIV Receiving Antiretroviral Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10002211; 002211-I
Record Dates: First submitted 2025-02-08; First posted 2025-02-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-15

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; ART intensification; Reservoir; lenacapavir; persistence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — lenacapavir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Participants will receive lenacapavir at 927 mg by subcutaneous injection (2x1.5 mL injections) on day 0 and 600 mg orally (2x300 mg tablets) on days 0 and 1, followed by 927 mg by subcutaneous injection (2x1.5 mL injections) at weeks 24 and 48.
  Interventions: Drug: Lenacapavir
- Standard of Care (No Intervention): Participants who are not randomized to lenacapavir will remain on their current ART regimens.

INTERVENTIONS:
Drug: Lenacapavir — Lenacapavir (Sunlenca) is a prescription drug approved by the Food and Drug Administration (FDA) for the treatment of people living with multidrug-resistant HIV. Lenacapavir is always used as part of a combination ART regimen. Participants will receive lenacapavir at 927 mg by subcutaneous injection (2x1.5 mL injections) on day 0 and 600 mg orally (2x300 mg tablets) on days 0 and 1, followed by 927 mg by subcutaneous injection (2x1.5 mL injections) at weeks 24 and 48.
  Arms: Interventional

SUMMARY:
Background:

Antiretroviral viral therapy (ART) allows people with human immunodeficiency (HIV) to live long, healthy lives. But ART is not a cure. HIV can remain in the body, in infected cells called reservoirs. If a person stops taking ART, the HIV can rebound and reach high levels in their blood. Researchers want to find ways to reduce the size of HIV reservoirs in people taking ART.

Objective:

To test a drug (lenacapavir) in people with HIV who are on effective ART. Lenacapavir, also called Sunlenca, is already approved for use in people with HIV who cannot be treated with standard ART.

Eligibility:

People aged 18 to 75 years with HIV that has been suppressed for at least 3 years with ART.

Design:

Participants will have 13 clinic visits over 2 years.

Participants will be screened. They will have a physical exam with blood tests. They will maintain their ART throughout the study.

Participants will undergo leukapheresis up to 6 times. Blood will be drawn via a tube in an arm. The blood will pass through a machine that separates out the white blood cells. The remaining blood will be returned to the body through a second tube.

Two-thirds of participants will take lenacapavir in addition to their regular ART. They will receive the drug as an injection under the skin 3 times at 6-month intervals. They will also take lenacapavir as 2 pills swallowed by mouth on the first 2 days of the study.

...

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

This is a treatment intensification study designed to ascertain the effects of lenacapavir intensification in people with HIV (PWH) with viral suppression on effective antiretroviral therapy (ART). Participants who fulfill the inclusion and exclusion criteria will be randomized in a 2:1 ratio to either continue their ART plus lenacapavir or continue their ART alone. Up to 24 participants will receive lenacapavir at 927 mg by subcutaneous (SC) injection (2x1.5 mL injections) on day 0 and 600 mg orally (2x300 mg tablets) on days 0 and 1, followed by 927 mg by subcutaneous injection (2x1.5 mL injections) at weeks 24 and 48. Participants in the lenacapavir arm will be followed for 48 weeks following the final injection. Up to 12 participants will remain on their prescribed ART regimens only. The size and rate of decay of intact HIV DNA reservoirs will be longitudinally monitored in each study group. All participants will undergo leukapheresis at baseline (prior to the first lenacapavir injection, if applicable) and at weeks 12, 24, 48, 72, and 96.

OBJECTIVES:

Primary Objective:

-To investigate the effect of the presence or absence of lenacapavir on intact HIV proviral DNA reservoirs in PWH who had been receiving virologically suppressive (<40 copies/mL) ART for greater than 3 years.

Secondary Objectives:

-To investigate the effect of the presence or absence of lenacapavir on residual plasma viremia (<40 copies/mL) in PWH who have been receiving virologically suppressive ART for greater than 3 years.

Exploratory Objectives:

* To investigate the effect of the presence or absence of lenacapavir on frequencies of CD4+ T cells carrying a) cell-associated HIV RNA, b) inducible HIV, and c) replication-competent virus.
* To investigate phenotypic changes on B, T, and natural killer cell markers.
* To investigate levels of HIV-specific T cells.
* To examine biomarkers in plasma.

ENDPOINTS:

Primary Endpoint:

-Changes in the intact HIV proviral reservoir size, measured by intact HIV proviral DNA assay (IPDA) in the blood CD4+ T-cell compartment from baseline to weeks 12, 24, 48, 72, and 96.

Secondary Endpoint:

-Changes in the residual HIV plasma viremia (1-39 copies/mL) from baseline to weeks 12, 24, 48, 72, and 96 (weeks 1, 2, 4, and 8 are optional).

Exploratory Endpoints:

* Frequencies of CD4+ T cells carrying cell-associated HIV RNA, inducible virion-associated HIV RNA, and replication-competent virus before, during, and after ART intensification with lenacapavir.
* Immunophenotyping of B, T, and natural killer cells using highdimensional flow cytometry before, during, and after ART intensification with lenacapavir.
* Measurements of the frequency of HIV-specific CD4+ and CD8+ T cells using overlapping HIV Gag peptides before, during, and after ART intensification with lenacapavir.
* Measurements of plasma biomarkers of immune activation and inflammation before, during, and after ART intensification with lenacapavir.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Able to provide informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Aged 18 years to 75 years.
4. In generally good health with an identified primary health care provider for medical management of HIV infection and willing to maintain a relationship with a primary health care provider while participating in the study.
5. Confirmed HIV-1 infection.
6. Total HIV DNA reservoir size greater than 300 copies/106 CD4+ T cells.
7. CD4+ T cell count >200 cells/mm^3 at screening.
8. Documentation of continuous ART treatment >3 years with suppression of plasma viral level below the limit of quantitation (<40 copies/mL). Individuals with <= 2 blips (>40 copies/mL) over 48 weeks prior to screening may be included provided they satisfy the following criteria:

   1. The blips are <=200 copies/mL.
   2. Succeeding viral levels return to below the limit of quantification (<40 copies/mL) on subsequent testing.
9. For individuals who can become pregnant (ie, participants who have not been postmenopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy), must have a negative pregnancy test at screening and within 48 hours prior to day 0. Participant-reported history is acceptable as documentation of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts, and vasectomy.
10. Participants who can become pregnant must agree to use 1 acceptable method of contraception when engaging in sexual activities that can result in pregnancy from 10 days prior to the first dose of lenacapavir through study follow up. Acceptable methods of contraception include the following:

    1. Contraceptive subdermal implant.
    2. Intrauterine device or intrauterine system.
    3. Combined estrogen and progestogen oral contraceptive.
    4. Injectable progestogen.
    5. Contraceptive vaginal ring.
    6. Percutaneous contraceptive patches.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of AIDS-defining illness within 3 years prior to enrollment.
2. History of systemic corticosteroids (eg, an equivalent dose of prednisone of >20 mg daily for >14 days), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy, or other medications considered significant by the principal investigator within the last 6 months.
3. Any clinically significant acute or chronic medical condition (eg, autoimmune diseases, cirrhosis, active malignancy that may require systemic chemotherapy or radiation therapy), other than HIV infection, that in the opinion of the investigator would preclude participation.
4. Hepatitis B or C infection as indicated by the presence of hepatitis B surface antigen or hepatitis C virus (HCV) RNA in blood.

   NOTE: Participants with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
5. Pregnancy or lactation.
6. Any licensed vaccine (eg, hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to the study enrollment.
7. Receipt of other investigational study agents within 28 days of enrollment and at any time during the study, including any experimental non-HIV vaccination within 2 weeks prior to enrollment.
8. Systemic immunosuppressive medications received within 3 months prior to enrollment. The following are not excluded:

   1. Corticosteroid nasal spray or inhaler.
   2. Topical corticosteroids for mild, uncomplicated dermatitis.
   3. Oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur (length of therapy 10 days, with completion in 30 days prior to enrollment).
   4. Cyclosporine eye drops
9. Active drug or alcohol abuse or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.
10. Laboratory abnormalities in the parameters listed below:

    1. Absolute neutrophil count <1,000 cells/mm^3
    2. Hemoglobin <10 g/dL
    3. Platelet count <100,000 cells/mm^3
    4. ALT >1.5 x ULN
    5. AST >1.5 x ULN
    6. Total bilirubin >1.5 x ULN
    7. Estimated glomerular filtration rate <30 mL/min/1.73m^2
11. Inability to undergo leukapheresis due to poor venous access or other medical conditions.
12. Concurrent treatment with any of the medications listed below:

    1. Antiarrhythmics: digoxin
    2. Anticoagulants: direct oral anticoagulants (DOACs), rivaroxaban, dabigatran, edoxaban
    3. Anticonvulsants: carbamazepine, oxcarbazepine, phenobarbital, phenytoin
    4. Antiretroviral Agents: atazanavir/cobicistat, atazanavir/ritonavir, efavirenz, nevirapine, tipranavir/ritonavir
    5. Antimycobacterials: Rifabutin, rifampin, rifapentine
    6. Corticosteroids (systemic): dexamethasone, hydrocortisone/cortisone
    7. Ergot derivatives: dihydroergotamine, ergotamine, methylergonovine
    8. Herbal products: St. John's wort c (Hypericum perforatum)
    9. HMG-CoA reductase inhibitors: lovastatin simvastatin
    10. Narcotic analgesics metabolized by CYP3A: fentanyl, oxycodone
    11. Tramadol
    12. Narcotic analgesic for treatment of opioid dependence: buprenorphine, methadone
    13. Opioid antagonist: naloxegol
    14. Phosphodiesterase-5 (PDE-5) inhibitors: sildenafil, tadalafil, vardenafil
    15. Sedatives/Hypnotics: midazolam (oral), triazolam
13. Past or current medical findings that are not listed above, which, in the opinion of the investigator, may pose additional risk from participation in the study, may interfere with the individual's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Co-enrollment guidelines: Co-enrollment in other trials or protocols involving apheresis is restricted, other than enrollment on observational studies. Co-enrollment in an interventional trial will require the approval of the principal investigator. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the principal investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Changes in the intact HIV proviral reservoir size, measured by IPDA in the blood CD4+ T-cell compartment from baseline to weeks 12, 24, 48, 72, and 96. | Through week 96.
  To compare the effect of the presence or absence of lenacapavir on intact HIV proviral DNA reservoirs in PWH who had been receiving virologically suppressive (<40 copies/mL) ART for greater than 3 years.

SECONDARY OUTCOMES:
Changes in the residual HIV plasma viremia (1-39 copies/mL) from baseline to weeks 12, 24, 48, 72, and 96 in the lenacapavir and control arm. | Through week 96.
  To compare the effect of the presence or absence of lenacapavir on residual plasma viremia (<40 copies/mL) in PWH who have been receiving virologically suppressive (<40 copies/mL) ART for greater than 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Yen C Lau, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with collaborators for analysis purposes. It will mostly be coded.
Time Frame: At the time of publication.
Access Criteria: Per repository and NIH Data Sharing requirements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002211-I.html